CLINICAL TRIAL: NCT00835315
Title: Prevalence of Psoriasis Alba in Psoriatic Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: hadassa medical organization,jerusalem,israel, hadassah medical organization
Other Study IDs: IPS001-HMO-CTIL
Record Dates: First submitted 2009-02-01; First posted 2009-02-03 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2009-02

CONDITIONS: Psoriasis
Keywords: interdigital psoriasis (psoriasis alba)
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 3: patients with psoriasis , patients with atopic dermatitis and healthy patients.

SUMMARY:
Interdigital psoriasis (psoriasis alba) is atypical and rare form of psoriasis that is often missed as it is commonly mistaken for either dermatoses or fungal infection.In this study we observed and analyzed the prevalence of psoriasis interdigital of palms and soles and brought medical awareness to dermatologists and family doctors this rare form of psoriasis. Thus, you can help to avoid mistaken diagnosis and the start of correct treatment as soon as possible.

DETAILED DESCRIPTION:
Hospitalized patients and outpatient clinic will be included in the study after receiving the signature of a inform consent.Patients groups : 100 patients with psoriasis,100 patients with atopic dermatitis and 100 healthy patients (control group).Patients with atopic dermatitis will be the secondary control group.Patients diagnosed with inflammatory condition of interdigital skin of the palms and soles will be checked by fungal microscopy test.If the fungal test is negative ,we need to prepare to a biopsy of the skin in this area .Following results of the skin biopsy conclusions can be shown about the prevalence of interdigital psoriasis in psoriatic patients enabling suitable treatment to be given to the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years old ,hebrew speakers, patients with psoriasis vulgaris or atopic dermatitis without systemic treatment

Exclusion Criteria:

* patients below 18 years old, pregnancy women, patients treated with systemic agents for psoriasis or atopic dermatitis(methotrexate,cyclosporin,neotigason)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients of dermatology depatment and outpatient clinic in the hospital
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-01

CONTACTS AND LOCATIONS:
Overall Officials: Vera Leibovici, MD, Principal Investigator — Hadassah Medical Organization; Natalya Lemster, MD, Principal Investigator — Hadassah Medical Organization